CLINICAL TRIAL: NCT03650764
Title: A Prospective Phase I and II Trial of Ramucirumab + Pembrolizumab in Patients With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Brief Title: Ramucirumab + Pembrolizumab in Patients With Recurrent/Metastatic Head and Neck Squamous Cell Carcinoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 201809094
Record Dates: First submitted 2018-08-27; First posted 2018-08-29 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Ramucirumab; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Phase I: Ramucirumab + Pembrolizumab (Experimental): -Ramucirumab will be administered IV over 1 hour on Day 1 of each 21-day cycle. Pembrolizumab will be administered as per standard of care (IV at a dose of 200 mg over 30 minutes on Day 1 of each 21-day cycle). On Day 1, pembrolizumab will be given after ramucirumab.
  Interventions: Drug: Ramucirumab; Drug: Pembrolizumab; Procedure: Peripheral blood
- Phase II: Ramucirumab + Pembrolizumab (Experimental): -Patients will be treated with ramucirumab at the RP2D on Day 1 and SOC pembrolizumab (200 mg IV over 30 minutes) on Day 1 of each 21-day cycle.
  Interventions: Drug: Ramucirumab; Drug: Pembrolizumab; Other: EORTC QLQ-30; Other: FACT H&N; Procedure: Peripheral blood

INTERVENTIONS:
Drug: Ramucirumab — Ramucirumab is an investigational agent for this trial and will be supplied by Lilly Oncology, free of charge to the patient
  Other Names: Cyramza
Drug: Pembrolizumab — Pembrolizumab is commercially available
  Other Names: Keytruda
Other: EORTC QLQ-30 — -Screening, start of cycle 2, start of cycle 5
  Arms: Phase II: Ramucirumab + Pembrolizumab
Other: FACT H&N — -Screening, start of cycle 2, start of cycle 5
  Arms: Phase II: Ramucirumab + Pembrolizumab
Procedure: Peripheral blood — -Baseline

SUMMARY:
The investigators hypothesize that inhibition of angiogenesis and PD-1 will be more effective than inhibition of PD-1 alone. The first step in pursuing proof of this hypothesis is to establish the safety and feasibility of combining ramucirumab with pembrolizumab, therefore the first part of this protocol is a de-escalation phase I trial of the combination of ramucirumab + pembrolizumab. The key objective of the phase I trial is to establish the safety and the recommended phase 2 dose (RP2D) of ramucirumab for this novel combination regimen in patients with recurrent/metastatic head and neck squamous cell carcinoma (RM-HNSCC). The second step in pursuing proof of this hypothesis is to establish the efficacy of ramucirumab (using the RP2D) with pembrolizumab. The second part of this protocol is a single arm phase II trial combining ramucirumab + pembrolizumab. The primary objective of the phase II trial is to determine the tumor response rates (complete response (CR) and partial response (PR)) of the treatment combination given as first line therapy in patients with RM-HNSCC.

ELIGIBILITY:
Inclusion Criteria:

* Incurable HNSCC, defined as RM disease not amenable to cure by surgery and/or radiation therapy or patient with HNSCC declines or is ineligible for curative therapy

  * In phase I, oral cavity, oropharynx, larynx, hypopharynx, nasopharynx, paranasal sinus, or salivary gland
  * In phase II, oral cavity, oropharynx, larynx, or hypopharynx
* Disease Evaluation:

  * In phase I, evaluable or measurable disease.
  * In phase II, measurable disease per RECIST 1.1
* Prior Treatment:

  * For phase I, any number of lines of prior therapy for RM-HNSCC.
  * For phase II, no prior systemic therapy for RM-HNSCC.
* At least 18 years of age.
* Performance status 0-2 (ECOG).
* Adequate blood and organ function as defined:

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Hemoglobin ≥ 9.0 g/dL
  * Total bilirubin ≤ 1.5 mg/dL
  * AST(SGOT) ≤ 3 x institutional upper limit of normal (IULN) and ALT(SGPT) ≤ 3 x IULN. In the setting of liver metastases, AST < 5 x IULN and ALT < 5 x IULN.
  * Creatinine ≤ 2 x ULN OR creatinine clearance ≥ 40 mL/min/1.73 m2
  * Urine protein to creatinine ratio (UPC) ≤ 1; if UPC ≥ 1, then a 24-hour urine protein must be assessed; patients must have a 24-hour urine protein value < 1 g to be eligible
  * INR ≤ 1.5 x ULN (≤ 3.0 x ULN if on anticoagulation) and PTT ≤ 1.5 x ULN (<3 x ULN if on anticoagulation) [Patients are allowed to be on anticoagulation]
* Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) beginning 14 days prior to first dose of ramucirumab, through the dosing period, and for at least 28 days after.
* Signed IRB approved written informed consent document.

Exclusion Criteria:

* Phase II: prior PD-1 inhibitor for treatment of incurable HNSCC. For phase I, prior PD-1 inhibitor therapy in the incurable setting is permitted.
* Radiation, chemotherapy, targeted or investigational therapy within 14 days of treatment start.
* Major surgery, presence of a non-healing, non-malignant ulcer within 14 days of treatment start; History of significant tumor site bleeding within 14 days of study consent.
* History of other malignancy ≤ 1 year previous with the exception of completely resected skin carcinoma or other cancers with a low risk of recurrence.
* Cirrhosis at a level of Child-Pugh B (or worse), Cirrhosis of any degree with a history of hepatic encephalopathy or clinically meaningful ascites (from cirrhosis requiring diuretics or paracentesis).
* Receiving any other investigational agents.
* Ongoing toxicity attributed to prior anti-cancer therapy that is > grade 1, except alopecia, anemia, fatigue or rash.
* Active central nervous system metastases: defined as currently receiving radiation therapy to metastatic CNS disease. Once radiation therapy is completed, patients with CNS disease are eligible if they meet all other criteria for enrollment.
* History of severe allergic reactions attributed to agents used in the study.
* Serious uncontrolled inter-current illness within the 3 months prior to study entry or psychiatric illness/social situations that would limit compliance with study requirements.
* Receiving systemic steroid therapy (in dosing exceeding 20 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of pembrolizumab.
* Has an active autoimmune disease (i.e. rheumatoid arthritis, lupus, Sjogren's syndrome) that has required IV or subcutaneous systemic treatment in the past 6 months (excluding rituxin). Replacement therapy (i.e. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of system treatment.
* GI perforation or fistula within 6 months of first dose of protocol therapy
* History of GI issues such as inflammatory bowel disease, ulcerative colitis, or Crohn's disease.
* Poorly controlled hypertension (defined as high blood pressure measurements [systolic blood pressures of ≥ 160 mmHg or diastolic blood pressures of > 100 mmHg] documented during the two-week interval prior to enrollment). Initiation or adjustment of antihypertensive medications to control blood pressure is permitted prior to study entry.
* Arterial thromboembolic events (including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina) within 3 months prior to first dose of treatment.
* GI Bleeding (grade 3 or 4) within 3 months prior to first dose.
* Pregnant and/or breastfeeding. Patient must have a negative serum pregnancy test within 7 days of first dose of treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2019-05-29 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Recommended phase 2 dose (RP2D) of ramucirumab combined with fixed dose pembrolizumab (Phase I patients only) | Completion of first cycle of treatment for all patients enrolled in Phase I portion of study (estimated to be 2.5 months)
  -The RP2D of ramucirumab is defined as the highest dose level at which fewer than 2 patients of a cohort of three patients experience a dose-limiting toxicity (DLT) during the first cycle.
Overall tumor response rate of ramucirumab and pembrolizumab (Phase II patients only) | Through 28 days after completion of treatment (estimated to be 6 months)
  * Overall tumor response rate = number of participants with complete response + partial response
  * Complete response (CR)=Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  * Partial response (PR)=At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

SECONDARY OUTCOMES:
Adverse event profile of the combination of ramucirumab and pembrolizumab (Phase I and II patients) as measured by the frequency of adverse events | Through 28 days after completion of treatment (estimated to be 6 months)
  -The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 will be utilized for all toxicity reporting.
Duration of overall response (Phase II patients only) | Through 28 days after completion of treatment (estimated to be 6 months)
  -Duration of overall response: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started).
  The duration of overall CR is measured from the time measurement criteria are first met for CR until the first date that progressive disease is objectively documented.
  -Duration of stable disease: Stable disease is measured from the start of the treatment until the criteria for progression are met, taking as reference the smallest measurements recorded since the treatment started, including the baseline measurements.
Progression-free survival (PFS) (Phase II patients only) | Through 28 days after completion of treatment (estimated to be 6 months)
  * PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.
  * Progressive disease: At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).
Overall survival (OS) (Phase II patients only) | Through 28 days after completion of treatment (estimated to be 6 months)
Changes in quality of life as measured by FACT H&N (Phase II patients only) | Baseline, start of cycle 2, and start of cycle 5 (estimated to be 12 weeks)
  * Median scores for each item and domain will be reported at each time point.
  * The general questionnaire, FACT-G, consists of 27 questions in four domains - physical (7), social/family (7), emotional (6), and functional (7). FACT-G is supplemented by a head and neck cancer specific subscale consisting of 11 questions to make up the 38 item FACT-H&N. Scores are calculated separately for each domain, and an unweighted summary score is calculated for the FACT-G and the total FACT H&N. The maximum score of 144 reflects the best possible quality of life
  * Answers to the questions range from 0=not at all to 4=very much
Changes in quality of life as measured by EORTC QLQ-C30 (Phase II patients only) | Baseline, start of cycle 2, and start of cycle 5 (estimated to be 12 weeks)
  * Median scores for each item and domain will be reported at each time point.
  * 30 items questionnaire with answers ranging from 1=not at all to 4=very much
  * includes five functional scales (physical, role, emotional, cognitive and social), three symptom scales (fatigue, nausea & vomiting and pain) and a global health status/QOL scale. Furthermore, it contains six single items (dyspnea, insomnia, appetite loss, constipation, diarrhea and financial difficulties)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas R Adkins, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Adkins D, Ley JC, Liu J, Oppelt P. Ramucirumab in combination with pembrolizumab for recurrent or metastatic head and neck squamous cell carcinoma: a single-centre, phase 1/2 trial. Lancet Oncol. 2024 Jul;25(7):888-900. doi: 10.1016/S1470-2045(24)00204-3. Epub 2024 Jun 5. PMID 38851207
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu